CLINICAL TRIAL: NCT01422265
Title: Patient Reported Symptoms in Ovarian Cancer
Brief Title: Patient Reported Symptoms in Ovarian Cancer (PRECISION)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28066; 130/070 (Other: Genentech)
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, observational, prospective study will include approximately 20 US-based centers, and approximately 142 patients diagnosed with epithelial ovarian cancer, primary peritoneal carcinoma or fallopian tube carcinoma, whose disease has recurred > 6 months after first-line platinum-based chemotherapy (first recurrence). Patients who have completed second-line chemotherapy and are currently in observation or undergoing bevacizumab maintenance treatment will be eligible to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented ovarian cancer, primary peritoneal carcinoma or fallopian tube carcinoma that has recurred > 6 months after platinum-based chemotherapy
* This must be the first recurrence of the epithelial ovarian cancer, primary peritoneal carcinoma or fallopian tube carcinoma
* Are at least two weeks but no more than 3 months after the completion of second-line cytotoxic chemotherapy
* Are currently under observation or being treated with bevacizumab as a second-line maintenance therapy
* Have a valid email address and access to the internet
* Provide voluntary written informed consent
* Speak and read English fluently

Exclusion Criteria:

* Current participation in a blinded clinical trial for ovarian cancer treatment. (Participation in a trial involving only supportive care medicines and/or growth factors is acceptable)
* Another primary diagnosis of cancer in a different site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with platinum-sensitive ovarian cancer in maintenance phase of second-line treatment
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in MD Anderson Symptom Inventory-Ovarian Cancer (MDASI-OC) sub-set symptom severity score before and after disease progression | Up to 9 months

SECONDARY OUTCOMES:
MDASI-OC Symptom Severity Score | Up to 9 months
MDASI-OC Symptom Interference Score | By month 9
HRQoL scores | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (30):
- United States (30):
  - Goodyear, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Salinas, California
  - Whittier, California
  - Englewood, Colorado
  - Farmington, Connecticut
  - New Britain, Connecticut
  - Augusta, Georgia
  - Hinsdale, Illinois
  - Joliet, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Missoula, Montana
  - Lincoln, Nebraska
  - Buffalo, New York
  - New York, New York
  - Watertown, New York
  - Canton, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Chattanooga, Tennessee
  - Salt Lake City, Utah
  - Annandale, Virginia
  - Tacoma, Washington